CLINICAL TRIAL: NCT06170099
Title: Assessment of Low Level Laser Therapy Effect on Treatment Outcomes of Bony Supported Distal Jet for Correction of Angle Class II Malocclusion (Randomized Clinical Trial)
Acronym: LLLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Rabab Abdel Hafez El Hosseini, MSD of Orthodontics, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-OR-19-01
Record Dates: First submitted 2023-11-29; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: This Study Focus on the Effect of Low-Level Light Therapy on the Amount of Upper Molar Distalization
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental)
  Interventions: Radiation: low level laser therapy; Device: bonny supported distal jet
- control group (Active Comparator)
  Interventions: Device: bonny supported distal jet

INTERVENTIONS:
Radiation: low level laser therapy — irradiation with LLLT by the following regimen 0, 3, 7 and 14 from the activation of the bony supported Distal Jet and then every 15 days till completion of distalization
  Arms: Laser group
Device: bonny supported distal jet — distal jet distalizing appliance is supported on two paramedian screw

SUMMARY:
The goal of this randomized clinical trial is to compare the effect of LLLT in adolescent patient with class II malocclusion. The main question it aims to answer is:

• is there a difference in the amount of distalization between laser and control groups? Participants will received bony supported distal jet. Researchers will compare laser group with control group to see if there is a difference in amount of distalization between groups.

DETAILED DESCRIPTION:
The aim of the present study is to assess the effect of low level laser therapy on treatment outcomes of bony supported distal jet for correction of 20 orthodontic patients with angle class II malocclusion. enrolled patient is randomly divided into 2 groups laser group and distal screw group. for result assessment dental casts and CBCT are taken before and after completion of distalization. both groups receives Distal Jet supported on 2 paramedian screw with laser therapy for laser group only.

ELIGIBILITY:
Inclusion Criteria:

* bilateral Angle's Class II malocclusion minimum of 1/4 cusp discrepancy, normal or low mandibular plane (MP) angle cases and no history of serious medical illness

Exclusion Criteria:

* subjects with skeletal Class II with retrusion mandibular profile, vertical growth pattern and steep mandibular plane angle and subjects with shallow or anterior open bite.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
amount of upper first molar distal movement | till achievement of class I molar relation, an average of 1 year
  mm/month

CONTACTS AND LOCATIONS:
Overall Officials: Rabab HF elhosseini, MSD, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar dental hospital, Cairo, Nasr City, Egypt